CLINICAL TRIAL: NCT04535843
Title: Precision Diagnosis and Prospective Cohort Study for Myasthenia Gravis: Multicenter Analysis in China
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Professor, Huashan Hospital
Other Study IDs: 2020-999
Record Dates: First submitted 2020-08-23; First posted 2020-09-02 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis; precision diagnosis; antibody detection
MeSH Terms: conditions — Myasthenia Gravis | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 1. Blood samples （Plasma/Serum/RNA/whole blood）
  2. Thymus/thymoma tissues obtained during thymic surgery
  3. Intercostal muscle specimens obtained during thymic surgery
  4. Lymph node samples obtained during thymic surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myasthenia gravis: 300 MG patients are anticipated for precision diagnosis and disease monitoring.
  Interventions: Other: Biomarkers and omics data

INTERVENTIONS:
Other: Biomarkers and omics data — To detect disease-related biomarkers and omics data, in this prospective MG cohort.

SUMMARY:
The present study is a prospective cohort study aiming to improve the clinical capacity in the diagnosis and natural history of Chinese patients with myasthenia gravis (MG). 300 MG patients are planned to recruit, document and prospectively follow up. Management of screening test and cohort manifestation are studied.

ELIGIBILITY:
Inclusion Criteria:

* fluctuating muscle weakness and fatigability, along with one of the below:
* more than 10% amplitude decrement in low frequency repetitive nerve stimulation,less than 10% amplitude increment in high frequency repetitive nerve stimulation;
* anti-AChR or MuSK antibody positivity;
* positive to the neostigmine test;
* understanding and assigning the informed consent form, and having a good compliance with the follow up.

Exclusion Criteria:

* excluding the possible diagnosis of Lambert-Eaton syndrome, congenital myasthenia syndrome,botulism injection, chronic progressive extraocular ophthalmoplegia, etc;
* poor compliance to the follow up.

Ages: 0 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from the outpatient clinics and inpatient wards are planned to be enrolled, as long as meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Myasthenia gravis foundation of America post intervention status | 3 years
  Myasthenia gravis foundation of America post intervention status (PIS) is assessed by the investigators during follow up. According to history inquiry and physical examination, participants are rated as clinical remission (no complain of myasthenia, no weakness at physical examination, and no therapies concerning MG for one year), pharmocological remission (no complain of myasthenia, no weakness at physical examination, but undertaking MG therapies at the last year), minimal manifestation (no complain of weakness, but showing weakness at physical examination), improvement (symptoms and signs), unchanged (symptoms and signs) , worsening(symptoms and signs), exacerbation(symptoms and signs), and death (medical record).

SECONDARY OUTCOMES:
Change From Baseline in Quantitative Myasthenia Gravis (QMG) Scores at the follow up | Baseline, 1 year, 2 year, and 3 year
  A quantitative MG scoring system (QMG Score) is essential in the objective evaluation of therapy for MG.This scoring system is based on quantitative testing of sentinel muscle groups. Total QMG score range from 0 (extreme disease severity) to 39 (none), higher score indicated less disease severity.
Change From Baseline in Activities of Daily Living (ADL) Scores at the follow up | Baseline, 1 year, 2 year, and 3 year
  The MG-ADL scale assesses the impact of MG on patients' daily functions. Physicians use this tool to score a patient's MG symptoms based on the patient's recall of symptoms during the prior week. A person's score can range from zero (normal) to 24 (most severe).
Change From Baseline in Myasthenia Gravis-Quality of Life Questionnaire-15 item (MG-QOL15) Scores at the follow up | Baseline, 1 year, 2 year, and 3 year
  The MG-QOL15 is helpful in informing the clinician about the patient's perception of the extent of and dissatisfaction with MG-related dysfunction. Total MG-QOL15 score range from 0 (none) to 60 (extreme disease severity), higher score indicated more disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, MD, Study Chair — Huashan Hospital, Shanghai,China
Locations (4):
- China (4):
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Obsterics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai

REFERENCES:
- [Derived] Jin L, Zou Z, Wang Q, Zeng W, Jiang Q, Chen J, Shi J, Yu Y, Hong D, Zeng Q, Tan S, Yue Y, Zhang Z, Zhang Y, Guo X, Du L, Zhao Z, Huang S, Chen Y, Wu Z, Yan C, Xi J, Song J, Luo S, Zhao C. Patterns and predictors of therapeutic response to efgartigimod in acetylcholine receptor-antibody generalized myasthenia gravis subtypes. Ther Adv Neurol Disord. 2025 Feb 18;18:17562864251319656. doi: 10.1177/17562864251319656. eCollection 2025. PMID 39974170
- [Derived] Jin L, He D, Zeng Q, Tan S, Shi J, Liu Y, Zou Z, Song J, Yan C, Huan X, Wang Y, Yang L, Xi J, Wu Z, Liu Z, Zheng J, Zhao C, Chu X, Luo S. Eculizumab in thymoma-associated myasthenia gravis: a real-world cohort study. Ther Adv Neurol Disord. 2024 Dec 25;17:17562864241309431. doi: 10.1177/17562864241309431. eCollection 2024. PMID 39735403